CLINICAL TRIAL: NCT07187128
Title: A Post-Market Study of Drug-Coated Peripheral Balloon Dilatation Catheter in Treating Femoropopliteal Artery Stenosis or Occlusive Lesions.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM-MK01
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Femoropopliteal Artery Stenoses or Occlusive Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VaSecure Drug-Coated Peripheral Balloon Dilatation Catheter (Experimental)
  Interventions: Device: drug coating balloon angioplasty

INTERVENTIONS:
Device: drug coating balloon angioplasty — The subjects underwent drug coating balloon angioplasty to treat femoropopliteal artery stenosis or occlusive lesions

SUMMARY:
T he Purpose of the Study is to evaluation of the Long-Term Safety and Effectiveness of a Drug-Coated Peripheral Balloon Dilatation Catheter in the Treatment of Femoropopliteal Artery Stenoses or Occlusive Lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 85 years, gender not restricted;
2. Rutherford grade 2 to 5
3. Target lesions located in the superficial femoral artery (SFA) and/or proximal popliteal artery requiring percutaneous transluminal angioplasty (PTA), with the following characteristics:

   * Diameter stenosis ≥70% by visual estimation or
   * Chronic total occlusion (CTO)
4. At least one native below-the-knee artery supplying the foot on the affected side preoperatively;
5. The guidewire can successfully pass through the target lesion site within the vascular lumen;
6. Agree to participate in this clinical study and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Absence of proximal inflow tract or persistent lack of proximal inflow after pretreatment
2. Type D or higher dissection occurring after target lesion predilation;
3. Residual diameter stenosis >50% following target lesion predilation;
4. Patients with known allergies to aspirin, clopidogrel, heparin, paclitaxel, contrast agents, etc.;
5. Abnormal function of vital organs (liver/kidney/brain) deemed unsuitable for intervention by investigators;
6. Documented allergy to aspirin, clopidogrel, heparin, paclitaxel/structural analogs, or contrast agents;
7. Patients currently undergoing dialysis or immunosuppressive therapy;
8. Presence of detectable thrombus in lower extremity arteries requiring intraoperative thrombolysis;
9. History of stroke or ST-elevation myocardial infarction within 6 months prior to procedure;
10. Pregnancy or lactation women;
11. Currently participation in other drug/medical device clinical trials without completion;
12. Patients deemed by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2028-10-10 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Patency Rate at 12 months post-procedure | 12 months
  12-month primary patency of the target lesion is defined as: absence of clinically driven target lesion revascularization and no Doppler ultrasound-diagnosed target lesion restenosis within 12 months postoperatively. Doppler ultrasound-diagnosed restenosis refers to a peak systolic velocity ratio (PSVR) ≥2.4 at the target lesion (indicating ≥50% luminal stenosis).
  Clinically Driven: Rutherford classification increase, ABI decrease, or imaging evidence of ≥70% stenosis.
  Target Lesion Revascularization: Includes any endovascular or open procedure at the target lesion site (e.g., PTA, stent placement, bypass surgery, thrombectomy, thrombolysis) or major amputation of the target limb.

SECONDARY OUTCOMES:
Device Success Rate | Immediately after procedure
Primary Patency Rate at 24 months post-procedure | 24 months
Target Lesion Revascularization (TLR) Rate at 12 amd 24 months post-procedure | 12 months; 24 months
Change in Rutherford classification from baseline at 6, 12, and 24 months postoperatively | 6, 12, 24 months
Change in ABI (ankle-brachial index) from baseline at 12 and 24 months postoperatively | 12, 24 months
MAEs Rates at 12 Months and 24 Months Post-Procedure | 12, 24 months
  MAEs: Include all-cause mortality within 30 days post-procedure, amputation of the treated limb, and clinically driven target vessel revascularization (TVR).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chognqing